CLINICAL TRIAL: NCT02056626
Title: Conditioned Pharmacotherapeutic Effects in Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, John Bisognano, M.D., Ph.D, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5R01HL105520 (NIH)
Record Dates: First submitted 2014-02-04; First posted 2014-02-06 (Estimated); Results first posted 2019-06-13 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Hypertension
Keywords: hypertension
MeSH Terms: conditions — Hypertension | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- arm 2 (Active Comparator): partial reinforcement, 6.25 mg twice daily, 25% of time (15 days)
  Interventions: Drug: carvedilol
- arm 3 (Active Comparator): controlled dosing schedule 6.25 mg twice daily (15 days)
  Interventions: Drug: carvedilol
- arm 4 (Active Comparator): controlled dosing schedule 6.25 mg twice daily, every other day (15 days)
  Interventions: Drug: carvedilol
- arm 1 (Active Comparator): standard therapy, 25 mg twice daily (15 days)
  Interventions: Drug: carvedilol

INTERVENTIONS:
Drug: carvedilol

SUMMARY:
The proposed research is designed to determine if the application of classical conditioning operations could influence the clinical effects of a regimen of antihypertensive drug therapy. It will be determined if, capitalizing on conditioned pharmacotherapeutic effects, patients can be effectively treated with smaller cumulative amounts of drug.

DETAILED DESCRIPTION:
The proposed research is designed to determine if the application of classical conditioning operations could influence the clinical effects of a regimen of antihypertensive drug therapy. In a double-blind, randomized, parallel-controlled clinical trial, It will be determined if, capitalizing on conditioned pharmacotherapeutic effects, patients can be effectively treated with smaller cumulative amounts of drug. To this end, some hypertensive patients will be treated on a partial rather than a continuous schedule of pharmacologic reinforcement. These patients will be compared to: (a) patients who continue to be treated under a standard regimen of pharmacotherapy at an effective dose of drug, and (b) patients who receive the same (reduced) cumulative amount of medication on a continuous schedule of reinforcement as that received by experimental patients treated under a partial schedule of reinforcement, and (c) patients who receive the same dose and frequency of carvedilol as the Partial Reinforcement Group but receive no intervening conditioned stimuli.

It is possible that a non-continuous schedule of pharmacologic reinforcement (and the concomitant reduced amount of active drug) will exert effects that are indistinguishable from a continuous (standard) regimen of pharmacotherapy (a higher cumulative amount of drug). That outcome or comparison, however, is not critical for evaluating the role of conditioning in the pharmacotherapy of hypertension. Specifically, we will test the hypotheses that:

1. patients treated under a partial schedule of antihypertensive medication will show a greater amelioration of symptoms than that achieved by patients treated with that same (reduced) amount of drug administered under a continuous schedule of reinforcement;

   Conditions permitting, we will also test the predictions that:
2. irrespective of initial treatment regimen, relapse will occur more quickly following withdrawal of active medication in patients who do not continue to receive conditioned stimuli (placebo) than in patients who continue to receive conditioned stimuli; and
3. when active drug is withdrawn and replaced by conditioned stimuli alone, resistance to extinction will be greater (i.e., rate of relapse will be less) among patients treated under a partial schedule of reinforcement than patients treated with the same amount of drug administered under a continuous schedule of reinforcement (the partial reinforcement effect).

Positive results would transform the study and practice of pharmacotherapy with respect to placebo effects by providing a new model within which to design treatment protocols for patients with chronic diseases that capitalizes on conditioned pharmacotherapeutic responses. The model, from which testable hypotheses can be derived, also provides a new framework for research on placebo effects and the mechanisms underlying such phenomena.

ELIGIBILITY:
Inclusion Criteria:

* systolic blood pressure between 140-160 mmHG
* between 18-80 years old

Exclusion Criteria:

* abnormal renal function
* currently pregnant, or trying to become pregnant
* being treated with a beta-blocker
* use of illicit drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-03; Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Bisognano, M.D., Ph.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] WOLF S. Effects of suggestion and conditioning on the action of chemical agents in human subjects; the pharmacology of placebos. J Clin Invest. 1950 Jan;29(1):100-9. doi: 10.1172/JCI102225. No abstract available. PMID 15399519
- [Background] LASAGNA L, MOSTELLER F, VON FELSINGER JM, BEECHER HK. A study of the placebo response. Am J Med. 1954 Jun;16(6):770-9. doi: 10.1016/0002-9343(54)90441-6. No abstract available. PMID 13158365
- [Background] KNOWLES JB. CONDITIONING AND THE PLACEBO EFFECT: THE EFFECTS OF DECAFFEINATED COFFEE ON SIMPLE REACTION TIME IN HABITUAL COFFEE DRINKERS. Behav Res Ther. 1963 Aug;1:151-7. doi: 10.1016/0005-7967(63)90018-4. No abstract available. PMID 14153340

RESULTS

PARTICIPANT FLOW:
Groups:
- Partial Reinforcement: partial reinforcement, 6.25 mg twice daily, 25% of time (15 days)
  carvedilol
- Controlled Dosing, Daily: controlled dosing schedule 6.25 mg twice daily (15 days)
  carvedilol
- Controlled Dosing, Every Other Day: controlled dosing schedule 6.25 mg twice daily, every other day (15 days)
  carvedilol
- Standard Therapy: standard therapy, 25 mg twice daily (15 days)
  carvedilol
Period: Overall Study
Arm/Group | Partial Reinforcement | Controlled Dosing, Daily | Controlled Dosing, Every Other Day | Standard Therapy
Started | 13 | 13 | 4 | 14
Completed | 10 | 12 | 4 | 14
Not Completed | 3 | 1 | 0 | 0
Not completed — patient did not follow directions | 3 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Partial Reinforcement | Controlled Dosing, Daily | Controlled Dosing, Every Other Day | Standard Therapy | Total
Number analyzed (Participants) | 13 | 13 | 4 | 14 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.62 (10.23) | 52.62 (12.14) | 58.00 (6.88) | 56.21 (5.70) | 51.89 (10.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 1 | 6 | 21
  Male | 5 | 7 | 3 | 8 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 2 | 1 | 2 | 10
  White | 5 | 10 | 2 | 12 | 29
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 1 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 4 | 14 | 44
Number of participants taking other antihypertensives [Count of Participants; unit: Participants] | 5 | 2 | 1 | 2 | 10
Mean systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 151.59 (7.22) | 152.64 (8.95) | 155.42 (9.62) | 151.88 (8.19) | 152.34 (8.05)

OUTCOME MEASURES:

1. Primary Outcome: Mean Systolic Blood Pressure
Time Frame: day 0
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Partial Reinforcement | Controlled Dosing, Daily | Controlled Dosing, Every Other Day | Standard Therapy
Number analyzed (Participants) | 10 | 12 | 4 | 14
mmHg | 151.59 (1.92) | 152.64 (2.38) | 155.42 (4.17) | 151.74 (2.05)

2. Primary Outcome: Mean Systolic Blood Pressure
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Partial Reinforcement | Controlled Dosing, Daily | Controlled Dosing, Every Other Day | Standard Therapy
Number analyzed (Participants) | 10 | 12 | 4 | 14
mmHg | 133.64 (2.58) | 132.92 (3.20) | 133.12 (3.20) | 135.00 (2.21)

3. Primary Outcome: Mean Systolic Blood Pressure
Time Frame: day 30
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Partial Reinforcement | Controlled Dosing, Daily | Controlled Dosing, Every Other Day | Standard Therapy
Number analyzed (Participants) | 10 | 12 | 4 | 14
mmHg | 138.90 (2.11) | 136.38 (3.34) | 139.27 (0.64) | 134.94 (2.71)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Partial Reinforcement | Controlled Dosing, Daily | Controlled Dosing, Every Other Day | Standard Therapy
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/4 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/4 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/4 | 0/14

LIMITATIONS AND CAVEATS:
This study was under enrolled and therefore not powered to answer the hypothesis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/26/NCT02056626/Prot_SAP_000.pdf
  • Informed Consent Form (2015-03-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT02056626/ICF_001.pdf